CLINICAL TRIAL: NCT00380055
Title: Reducing Cancer Disparities for American Indians in the Rural Intermountain West
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sletten Cancer Institute (Other); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Randall W. Rupper, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18388; 1A0CMS300067
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer; Colorectal Cancer; Breast Cancer; Cervical Cancer; Lung Cancer
Keywords: Cancer Screening; Navigators; Community Outreach; Behavioral Change; Access
MeSH Terms: conditions — Prostatic Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Screening Navigation (Experimental): Individuals without a study cancer who receive services of a navigator.
  Interventions: Behavioral: Navigation Services
- Treatment Navigation (Experimental): Individuals with a study cancer who receive navigation services.
  Interventions: Behavioral: Navigation Services
- Screening Education (Active Comparator): Rather than receiving navigation, these participants receive general cancer education appropriate to Medicare enrollees.
  Interventions: Behavioral: Cancer education
- Treatment Education (Active Comparator): Rather than receiving navigation services, these participants receive cancer education appropriate to Medicare recipients.
  Interventions: Behavioral: Cancer education

INTERVENTIONS:
Behavioral: Navigation Services — Navigators (community health workers) identify and assist in overcoming barriers to appropriate cancer care.
  Arms: Screening Navigation; Treatment Navigation
Behavioral: Cancer education — Community health workers provide cancer education appropriate for Medicare participants.
  Arms: Screening Education; Treatment Education

SUMMARY:
The purpose of this demonstration is to evaluate the effectiveness of using community outreach workers (navigators) to help American Indians living in rural areas overcome barriers to appropriate cancer screening, diagnosis, and treatment.

DETAILED DESCRIPTION:
Even for American Indians who have coverage with Medicare, disparities have been noted in the provision of cancer screening, diagnosis, and treatment. These disparities have been related to a variety of health-system, health-financing, geographic, and cultural barriers. We hypothesize that the use of lay community outreach workers will be an effective means of identifying and overcoming these barriers in order to improve the proportion of Medicare-eligible American Indians who receive recommended screening and diagnosis for prostate, breast, colon, and cervical cancer, and the proportion of individuals receiving appropriate treatment for prostate, breast, colon, cervical, and lung cancer. Community clusters randomized to this form of cancer navigation will be compared with community clusters randomized to receive educational outreach only.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Medicare Part B
* Self-reported American Indian

Exclusion Criteria:

* Have cancer other than study cancer
* Medicare Part C enrolled

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals receiving recommended screening for prostate, breast, colorectal, and cervical cancer. | four years

SECONDARY OUTCOMES:
Proportion of individuals receiving recommended diagnostic follow-up for prostate, breast, colorectal, and cervical cancer. | four years
Proportion of individuals receiving recommended treatment for prostate, breast, colorectal, cervical, and lung cancer. | four years
Cost-effectiveness of using community navigators to improve cancer care among rural Native Americans. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall W. Burt, MD, Principal Investigator — Huntsman Cancer Institute
Locations (2):
- United States (2):
  - Sletten Cancer Institute, Great Falls, Montana
  - Huntsman Cancer Institute, Salt Lake City, Utah